CLINICAL TRIAL: NCT04884230
Title: Oversewing Staple Line of the Gastric Remnant in Gastric Bypass Reduces Postoperative Bleeding.
Brief Title: Oversewing Staple Line of The Gastric Remnant
Status: Completed | Type: Observational
Sponsor: Unidad Internacional de Cirugia Bariatrica y Metabolica (Other)
Responsible Party: Principal Investigator, Andres Maldonado, Dr., Unidad Internacional de Cirugia Bariatrica y Metabolica
Other Study IDs: UnidadInternacional
Record Dates: First submitted 2021-05-03; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Gastric Bypass; Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: We selected 225 patients (group A) from the period 2019-2020 where the stapling line of the gastric remnant was oversewn and another group of 225 patients (group B) from the period of 2017-2018 with stapling alone.
  Interventions: Procedure: Oversewing
- Group B: We selected 225 patients (group A) from the period 2019-2020 where the stapling line of the gastric remnant was oversewn and another group of 225 patients (group B) from the period of 2017-2018 with stapling alone.

INTERVENTIONS:
Procedure: Oversewing — Oversewing of the gastric remnant
  Groups: Group A

SUMMARY:
Background: Roux-en-Y gastric bypass (RYGB) is a surgery with low rate complications. However, it is not exempt from them, and 1-6% suffer complications such as postoperative bleeding. Many intraoperative techniques have been evaluated to reduce postoperative bleeding, like the oversewing or reinforcement of the staple line. This study aims to evaluate the rate of postoperative bleeding in the oversewing of the staple line of the gastric remnant group versus the stapling only group.

Methods: This is a 2-center, case-control study. The investigators randomly selected two groups who underwent RYGB or OAGB: group A (n=225) with oversewing from 2019-2020 and group B (n=225) with stapling only between the period of 2017-2018; both groups with similar demographic characteristics.

DETAILED DESCRIPTION:
This case-control study was conducted in the International Unit of Bariatric and Metabolic Surgery of "Clinica La Sagrada Familia" located in Maracaibo, Venezuela, and in "Grupo Medico Santa Paula" Caracas, Venezuela. All procedures were performed by a single experienced bariatric surgeon during the period 2017-2020. The Ethics committees of Clinica "La Sagrada Familia" and "Grupo Medico Santa Paula" approved this study. The investigators selected 225 patients (group A) from the period 2019-2020 where the stapling line of the gastric remnant was oversewn and another group of 225 patients (group B) from the period of 2017-2018 with stapling alone.

ELIGIBILITY:
Inclusion Criteria:

* Our inclusion criteria were patients older than 18 years, body mass index (BMI) > 30kg/m2 with or without comorbidities that underwent RYGB or one anastomosis gastric bypass (OAGB).

Exclusion Criteria:

* We exclude from our study any patient with psychiatric disorder, open surgery history, history of previous bariatric surgery, non-controlled comorbidity at the moment of surgery, and patients under the age of 18

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients older than 18 years, body mass index (BMI) > 30kg/m2 with or without comorbidities that underwent RYGB or one anastomosis gastric bypass (OAGB).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2017-02-05 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Reduce bleeding | Through study completion, 6 month average
  assessing melena

CONTACTS AND LOCATIONS:
Locations (1):
- CCSF, Maracaibo, Zulia, Venezuela

IPD SHARING:
Plan to Share IPD: No
Personal.